CLINICAL TRIAL: NCT05706740
Title: Understanding Patterns of Deprescribing Antithrombotic Medication During End-of-Life Care in Cancer Patients Across the European Union
Brief Title: Towards Cancer Patient Empowerment for Optimal Use of Antithrombotic Therapy at the End of Life
Acronym: SERENITY
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Prof. Stavros Konstantinides, MD, Coordinating Investigator, Johannes Gutenberg University Mainz
Other Study IDs: CTH C012
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Terminal Cancer
Keywords: palliative care; antithrombotic therapy; deprescription; advanced cancer; thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Physician survey on antithrombotic medication during end-of-life care in cancer patients — Participating healthcare professionals will be asked to complete the survey electronically within seven days. The survey will consist of general questions (i.e., "Have you ever considered deprescribing antithrombotic medicine"?), a discrete choice experiment (DCE), and questions involving actual decision-making in patients.
  For the DCE, participants will be presented a sequence of choice sets with (hypothetical) scenarios that vary along several characteristics (attributes; e.g., bleeding risk, thrombotic risk). Attributes will be further specified by varying choice levels (attribute levels; e.g., low or high bleeding risk). Participants will be asked to select the healthcare intervention with the highest benefit for the patient according to their opinion.
  Finally, participants will be asked to describe actual decisions they made in max. three consecutive patients with active cancer, who were considered to receive end-of-life care.

SUMMARY:
Despite the fact that antithrombotic therapy (ATT) has little or even negative effects on the well-being of cancer patients during their last year of life, stopping ATT is rare in clinical practice. In contrast, antithrombotic therapy is often continued until death, resulting in excess bleeding, higher healthcare costs, and increased disease burden. SERENITY aims to develop an information-driven, palliative care shared decision-making process enabled by a user-friendly, easily accessible, web-based shared-decision support tool (SDST) that will facilitate treatment decisions regarding appropriate use of antithrombotic therapy in cancer patients at the end of life. SERENITY will use a comprehensive approach consisting of a combination of realist review, flash mob research, qualitative interviews, epidemiologic studies, and a randomized controlled trial.

The sub-project described here uses the flashmob research approach to address healthcare professionals from various institutions, who deal with end-of-life care in cancer patients, or prescribe antithrombotic medication to cancer patients.The survey will be conducted with approx. 800 physicians from eight European countries, all represented in the SERENITY consortium.

DETAILED DESCRIPTION:
Deprescribing is an important part of palliative care to prevent polypharmacy, which is associated with increased risk of adverse drug events, drug-drug and drug-disease interactions, reduced functional capacity, multiple geriatric syndromes, medication nonadherence, and higher healthcare costs. One of the most widely used cardiovascular drug classes in cancer patients in a palliative setting are antithrombotics, including anticoagulant and anti-platelet substances. Antithrombotic drugs, e.g., direct oral anticoagulants (DOACs), low-molecular-weight heparins (LMWH), vitamin-K antagonists (VKA) and so-called antiplatelet agents (such as acetyl salicylic acid and P2Y12 inhibitors), are indicated in patients with prosthetic heart valves, in those with venous thromboembolism (VTE) or pulmonary embolism (PE), for stroke prevention in atrial fibrillation as well as in patients with established atherosclerotic cardiovascular disease (such as myocardial infarction, stroke, or peripheral artery disease). Most patients have been receiving these drugs chronically before their cancer was diagnosed, while others are prescribed them in order to treat or prevent cancer-associated thrombosis. Obviously, decisions on deprescribing antithrombotics heavily depend on the indication of the antithrombotic drug in addition to patient and healthcare professional preferences and experience, and on the estimated life expectancy of the patient.

Understanding current patterns of management of antithrombotic therapy as well as the rationale and preferences behind these patterns is crucial for improving clinical practice. Since deprescribing patterns and rationale may largely differ across the European Union, relevant data at a large scale is needed to fully understand and appreciate the relevant decision processes.

The insights gained in this study are a first step towards the development of a clinical decision tool supporting decisions on antithrombotic therapy in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Healthcare professionals from various institutions, who deal with end-of-life care in cancer patients, or prescribe antithrombotic medication to cancer patients

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare professionals to be recruited will involve general practitioners, palliative care specialists, nursing home physicians, geriatrists, vascular medicine physicians, oncologists, haematologists, pulmonologists, cardiologists, neurologists, and vascular surgeons with equal gender representation and distribution of experienced versus less experienced (young professionals) physicians.
  The survey will be conducted in 8 European countries (Denmark, France, Germany, Italy, The Netherlands, Poland, Spain, United Kingdom).
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2023-02-28 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Current practice patterns across Europe with regard to the use of antithrombotic treatment in end-of-life care of cancer patients | 7 days
  The main analysis of the FMR will be descriptive. Responses to the Discrete Choice Experiments will be used to generate preference coefficients for each level (e.g., high/low) of each attribute (e.g., bleeding risk)
Relevance of patient's age for the decision on continuation or discontinuation of antithrombotic therapyin cancer patients during end-of-life care | 7 days
Relevance of patient's prognosis for the decision on continuation or discontinuation of antithrombotic therapyin cancer patients during end-of-life care | 7 days
Relevance of patient's performance status (Eastern Cooperative Oncology Group | 7 days
  (ECOG)) for the decision on continuation or discontinuation of antithrombotic therapy
Relevance of patient's type of antithrombotic medication for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of patient's indication for antithrombotic medication for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of patient's thrombotic risk for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of patient's bleeding risk for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of patient's symptom burden for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of patient's medication burden for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of patient's preference (pro/contra continuation) for the decision on continuation or discontinuation of antithrombotic therapy | 7 days
Relevance of physician's experience (with deprescribing) for antithrombotic medication for the decision on continuation or discontinuation of antithrombotic therapy | 7 days

CONTACTS AND LOCATIONS:
Locations (12):
- Aalborg University Hospital, Aalborg, Denmark
- France (2):
  - Assistance Publique - Hôpitaux de Paris, Paris
  - Centre Hospitalier Universitaire Saint Etienne, Saint-Etienne
- Universitaetsmedizin Der Johannes Gutenberg-Universitaet Mainz, Mainz, Germany
- Società Per L'Assistenza Al Malato Oncologico Terminale Onlus, Ragusa, Italy
- Netherlands (3):
  - Academisch Ziekenhuis Leiden (Lumc), Leiden
  - Erasmus Universitair Medisch Centrum Rotterdam, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Centrum Medyczne Ksztalcenia Podyplomowego, Warsaw, Poland
- Fundació Clínic Per A La Recerca Biomèdica, Barcelona, Spain
- United Kingdom (2):
  - Cardiff University, Cardiff
  - University of Hull, Hull

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT05706740/Prot_SAP_000.pdf